CLINICAL TRIAL: NCT03389334
Title: Effects of Myofascial Release Massage on Pain Levels, Range of Motion, and Muscle Strength in Unilateral Lower Limb Amputees
Brief Title: Massage on Pain Levels, Range of Motion, and Muscle Strength in Unilateral Lower Limb Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Heather Appling, Assistant Professor Department of Orthotics and Prosthetics, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5170458
Record Dates: First submitted 2017-12-13; First posted 2018-01-03 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Amputation
MeSH Terms: interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- massage group (Experimental): Subjects will complete the SF-36, ODI, demographics surveys and then will receive pre-treatment range of motion, muscle strength and visual analogue pain scale prior to massage. Then will have a 45-minute myofascial release massage. Then they will fill out the visual analogue pain scale again. (Approximately 90-minutes) The second and third visits: visual analogue scale prior to the treatment; 45-minute massage, by the same therapist who treated them during the initial visit, and will fill out a second visual analog pain scale following the treatment. (Approximately 60-minutes) The fourth visit: visual analogue pain scale and 45-minute massage; post-treatment SF-36, ODI surveys, visual analogue pain scale, post-treatment range of motion and muscle strength.
  Interventions: Other: massage

INTERVENTIONS:
Other: massage — The techniques include myofascial release and manual active and passive stretching with the intention to lengthen overly contracted or shortened tissue, increase range of motion, and restore any malpositioning of structural landmarks as defined by its contralateral counterpart. By addressing the symptoms of the somatic dysfunction, you will in turn reduce the overall perceived pain in the body caused in these related tissues. The duration of each massage treatment session will be 45 minutes long and therapists will use a timer to ensure all subjects receive the same length of treatment. Patients will continue to receive treatment from the same therapist to maintain consistency of results.

SUMMARY:
The purpose of this graduate research study is to explore the therapeutic benefits of Myofascial Release massage on lower limb amputees with pain levels, range of motion, and muscle strength.

DETAILED DESCRIPTION:
There are no other studies that address the effects of massage therapy as a treatment option for lower limb amputees suffering from lower back pain or the effects this has on muscle performance and/or range of motion. In addressing the physical, psychological, and social needs of a person living with limb loss, there should be a consideration for a multidisciplinary approach that could potentially include massage therapy as a fundamental standard of care. Therefore, the purpose of this graduate student research study is to test whether myofascial release massage can improve lower back pain levels in lower limb amputees and consequently improve quality of life and other measurable variables such as range of motion and muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Pain in the lower back region
* Trans-tibial, trans-femoral, knee disarticulation, or Symes amputees
* Unilateral lower limb amputation
* Subject willing to receive massage once a week over a 4 week span
* Subject must be willing to abstain from over-the-counter and prescription pain medication 24 hours before each treatment

Exclusion Criteria:

* Open wounds within the treatment area
* Bilateral lower limb amputees
* Pregnant subjects (self-reported)
* Lymphedema
* Amputation distal to ankle
* Subjects who currently receive regular massage treatments
* Subjects taking anticoagulant medication
* Subjects with allergies to coconut oil

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-06-16 (Actual); Study Completion 2018-06-16 (Actual)

PRIMARY OUTCOMES:
Low Back Pain | Change in low back pain between baseline and study completion at the fourth week (Visit 4).
  Subject's lower back pain data will be collected through the Owestry Disability Index (ODI). It is valid and reliable in a variety of settings . Patients select statements that are most applicable to their current situation in the following areas: intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function (if applicable), ability to stand, social life, sleep quality, and ability to travel. The questionnaire will take less than 5 minutes. Questionnaire is given at the beginning of the study and then will be compared with the responses after the 4 week treatment.
visual analog pain scale | Change in visual analog pain scale score between baseline and study completion at the fourth week (Visit 4).
  A Visual Analog Scale, consisting of a 10 cm long horizontal line which represents various levels of pain with "No Pain" at one end and "Unbearable Pain" at the other will be given.

SECONDARY OUTCOMES:
Range of Motion | Change in range of motion as measured by goniometer between baseline and study completion at the fourth week (Visit 4).
  In order to determine whether subjects had any improvement in their range of motion (ROM) investigators will measure their hip and knee joint (if applicable). Investigators will use a standard 12 inch plastic goniometer to measure and record the angles at each joint. The specific goniometer was manufactured by Ever Ready First Aid Medical Supply Corp. in Brooklyn, NY. This tool can measure up to 360 degrees in 1 degree increments and has been calibrated according to the International Standards of Measurement.
Muscle strength | Change in muscle strength score as measured by the MMT between baseline and study completion at the fourth week (Visit 4).
  Regarding muscle strength, investigators will perform a Manual Muscle Test (MMT) according to the 9th edition of Daniels & Worthington's Muscle Testing. The specific techniques described in this text focus the MMT on joint movements rather than individual muscles (for example knee extension vs. rectus femoris). The most common procedure is called the break test, in which the limb is placed and held at the end of the available range (for one-joint muscles) or at mid-range (for two-joint muscles) and manual resistance is applied by the therapist in the direction of the line of pull of the muscle(s) being tested. A numerical and qualitative score is then assigned to the muscle(s) ranging from 5: Normal (N) to 0: No activity (0).

CONTACTS AND LOCATIONS:
Overall Officials: Heather Appling, MSOP, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda Universtiy, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No